CLINICAL TRIAL: NCT06492135
Title: Safety, Tolerability and Pharmacokinetics Study of Multiple Rising Subcutaneous Doses of Survodutide in Chinese Participants With Overweight or Obesity (BMI 24.0 to 40.0 kg/m2) (Non-randomization, Open Label, Parallel Group Design)
Brief Title: A Study in Chinese People With Overweight or Obesity to Test How Different Doses of Survodutide Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0013
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Participants with a body mass index (BMI) ranging from ≥27.0 kg/m² to ≤40.0 kg/m² (Experimental)
  Interventions: Drug: survodutide
- Arm 2: Participants with a body mass index (BMI) ranging from ≥24.0 kg/m² to <27.0 kg/m² (Experimental)
  Interventions: Drug: survodutide

INTERVENTIONS:
Drug: survodutide — survodutide

SUMMARY:
This study is open to Chinese adults aged 18 to 60 with overweight or obesity. People can join the study if they have a Body Mass Index from 24 to 40.0 kg/m2.

Survodutide is a medicine being developed to help people with overweight or obesity. The purpose of this study is to find out how different doses of survodutide are taken up in the body. Other goals are to test if participants can tolerate different doses of survodutide and whether survodutide helps people with overweight or obesity.

Participants receive survodutide as an injection under the skin once a week for 7.5 months. During this time, participants visit the study site 33 times. 4 of the visits require a stay in the hospital. At the visits, doctors take blood samples to measure the levels of survodutide in participants' blood. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Age of 18 to 60 years
* 40≥ body mass index (BMI) ≥30 kilogram (kg)/ square meters (m²) at screening, or 30> BMI ≥27 kg/m² at screening with the presence of at least one of the following weight-related complications

  * Hypertension
  * Dyslipidemia
  * Obstructive sleep apnea
  * Cardiovascular disease (CVD) (e.g. heart failure (HF) with New York Heart Association (NYHA) functional class II-III, history of ischemic or hemorrhagic stroke or cerebrovascular revascularization procedure [e.g. carotid endarterectomy and/or stent], myocardial infarction (MI), coronary artery disease, or peripheral vascular disease)
  * Non-alcoholic steato hepatitis (NASH), as assessed in medical records by histological liver assessment (within the last 6 months) or overweight but otherwise healthy participants with BMI ≥ 24 but < 27 kg/m² according to the assessment of the investigator, based on a complete medical history, physical examination, vital signs (BP, PR), 12-lead electrocardiogram (ECG), and clinical laboratory tests at screening.
* stable body weight in the 3 months prior to screening visit (defined as no more than 5% change by self-report)
* further inclusion criteria apply

Exclusion Criteria:

* Repeated measurement of sitting blood pressure (BP) ≥160/95 millimeter of mercury (mmHg), or pulse rate (PR) >100 beats per minute (bpm) after 5 minutes of resting at screening visit.
* Exposure to any glucagon-like-peptide 1 receptor (GLP-1R) agonist (including combination products) within three months prior to screening visit, or any previous exposure to survodutide, or history of relevant allergy or hypersensitivity (including allergy intolerability or lack of efficacy to trial medication or drugs that belongs to the GLP-1R agonist class).
* Trial participants with the following laboratory findings at screening are excluded:

  * Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) elevation ≥3× upper limit of normal (ULN)
  * Total bilirubin ≥1.2× ULN
  * Calcitonin ≥100 picograms per milliliter (pg/mL) (29.26 picomoles per litre (pmol/L))
  * Glycosylated hemoglobin A1c (N-(1-deoxy)-fructosyl-hemoglobin) (HbA1c) > upper limit of normal (ULN)
* History of either chronic or acute pancreatitis or elevation of serum lipase or amylase >2x ULN as measured by the laboratory at screening
* further exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
AUC0-168 (area under the concentration-time curve of survodutide in plasma over the time interval from 0 to 168h) | up to 7 days
Cmax (maximum measured concentration of survodutide in plasma) after the first dose | up to 7 days
Cmax (maximum measured concentration of survodutide in plasma) after multiple doses | up to 7 days

SECONDARY OUTCOMES:
Percentage (%) of participants withdrawn due to adverse events from up-titration by dose | up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Central Hospital of Xuhui District, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com